CLINICAL TRIAL: NCT04344158
Title: A Randomized, Controlled, Open-label, Multicenter Phase III Clinical Trial of AK105 Injection Combined With Anlotinib Hydrochloride Capsules Versus Sorafenib in Subjects With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Phase III Clinical Trial of AK105 Injection Combined With Anlotinib Hydrochloride Capsules Versus Sorafenib in Subjects With Advanced Hepatocellular Carcinoma (HCC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AK105-III-02
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK105 combined with Anlotinib (Experimental): AK105 200mg intravenously (IV) on day 1 of each 21-day cycle plus Anlotinib capsules 10mg given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: AK105 Injection; Drug: Anlotinib Hydrochloride Capsules
- Sorafenib Tosylate Tablets (Active Comparator): Sorafenib Tosylate Tablets 400mg given orally, twice daily in 21-day cycle.
  Interventions: Drug: Sorafenib Tosylate Tablets

INTERVENTIONS:
Drug: AK105 Injection — AK105 200mg intravenously (IV) on day 1 of each 21-day cycle.
  Arms: AK105 combined with Anlotinib
Drug: Anlotinib Hydrochloride Capsules — Anlotinib capsules 10mg given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Arms: AK105 combined with Anlotinib
Drug: Sorafenib Tosylate Tablets — Sorafenib Tosylate Tablets 400mg given orally, twice daily in 21-day cycle.
  Arms: Sorafenib Tosylate Tablets

SUMMARY:
This is a randomized, controlled, open-label, multicenter study to evaluate efficacy of AK105 injection combined with Anlotinib Hydrochloride Capsules versus Sorafenib. Patients are treated with AK105 injection combined with Anlotinib Hydrochloride Capsules or Sorafenib, with 2:1 random ratio. Every 21 days is a treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-75 years old; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.

  2. Histopathology or cytology confirmed as HCC. 3. Has not received any systematic treatment for HCC. 4. Stage B or C in the Barcelona Clinic Liver Cancer (BCLC) classification, and is not suitable for surgery or local treatment, or progress after surgery or local treatment.

  5. Child-Pugh liver function classification : A or B (≤7 points). 6. Central nervous system metastasis has no clinical symptoms or is stable at least 4 weeks after treatment.

  7. Quantification of HBV DNA <500IU/ml or 2500 Copys/ml, and anti-HBV therapy should be given for at least 2 weeks before the first administration; Quantification of HCV RNA is positive must complete antiviral therapy at least 1 month before the first administration.

  8. Patients who progress after local treatment should be at least 4 weeks after the end of local treatment.

  9. Radiotherapy for bone metastases accompanied by clinical symptoms must be completed at least 2 weeks before the first administration.

  10. Has at least one measurable lesion. 11. Adequate organ function. 12. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

  13.Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Histopathology or cytology confirmed as fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, hepatobiliary cell carcinoma, mixed liver cancer, etc.

  2. Has used anti-angiogenic drugs such as anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, bevacizumab, or related immunotherapy drugs for PD-1, PD-L1, etc.

  3. Has received systemic treatment such as chemotherapy and biological therapy. 4. Has a history of hepatic encephalopathy. 5. According to imaging examination, the portal vein has invasion of cancer embolus, inferior vena cava or heart involvement.

  6. Hepatitis B with hepatitis C or hepatitis D infection. 7. Has received or planned to receive organ transplantation. 8. Has other malignant tumors within 5 years. 9. Has multiple factors affecting oral medication. 10. Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

  11. Has any bleeding or bleeding events ≥grade 3 in the first 4 weeks before the first administration.

  12. Has unhealed wounds, fractures, active gastric and duodenal ulcers, positive continuous fecal occult blood, ulcerative colitis in the first 4 weeks before the first administration.

  13. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  14. Has received surgery, or unhealed wounds within 4 weeks before the first administration.

  15. Has drug abuse history that unable to abstain from or mental disorders. 16. Has any serious and / or uncontrolled disease. 17. Has received vaccination or attenuated vaccine within 4 weeks prior to the first administration.

  18. Has received anti-tumor Traditional Chinese Medicine within 2 weeks before the first administration.

  19. Severe hypersensitivity after administration of other monoclonal antibodies.

  20. Has any active autoimmune disease or history of autoimmune disease. 21.Immunosuppressant or systemic or absorbable local hormone therapy is required to achieve the aim of immunosuppression (dose > 10mg/ day prednisone or other therapeutic hormones) and is still used within 2 weeks after the first administration.

  22.Has participated in other anticancer drug clinical trials within 4 weeks. 23.Portal hypertension with high risk of hemorrhage, or have red sign confirmed by gastroscopy.

  24.According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 96 weeks
  OS defined as the time from the first dose to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall response rate（ORR） | Up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | Up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | Up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (81):
- China (81):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Ditan Hospital.Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital.Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital.Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The first hospital of Lanzhou University, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital，Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Nanning People's Hospital, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical Universit, Haikou, Hainan
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - First Hospital Of Qinhuangdao, Qinhuangdao, Hebie
  - Affiliated Hospital of Chengde Medical University, Chengde, Heibei
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang First People's Hospita, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Xinxiang central hospital, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancar Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan Cancer Hospital(Department II of Gastroenterology and Urology/Hepatobiliary Surgery), Changsha, Hunan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital Affiliated to Jilin Universit, Changchun, Jilin
  - Jilin Guowen Hospital, Changchun, Jilin
  - Gansu Provincial Hospital, Gansu, Lanzhou
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The Sixth People's Hospital Of Shenyang, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Baoji Central Hospital, Baoji, Shaanxi
  - Hanzhong Central Hospital, Hanzhong, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng people's Hospital, Liaocheng, Shandong
  - Yidu Central Hospital Of Weifang, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fuadn University, Shanghai, Shanghai Municipality
  - The Third Affiliated Hospital of the Second Military Medical University of the Chinese people's Liberation Army, Shanghai, Shanghai Municipality
  - Shanxi Provinaial Cancer Hospital, Taiyuan, Shanxi
  - Tangdu Hospital of the Fourth Military Medical University of the People's Liberation Army of China, Xi’an, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shanxi Provincial Cancer Hospital, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Affiliated Hospital of Chengdu University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University Cancar institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - Shulan (Hangzhou) hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Zhou J, Bai L, Luo J, Bai Y, Pan Y, Yang X, Gao Y, Shi R, Zhang W, Zheng J, Hua X, Xu A, Hu S, Zhang F, Yang X, Da M, Wang R, Ma J, Jia W, Quan D, Peng C, Yang W, Yin G, Qi Y, Zhang G, Du X, Mao X, Meng Z, Jiao S, Fan J; APOLLO Study Group. Anlotinib plus penpulimab versus sorafenib in the first-line treatment of unresectable hepatocellular carcinoma (APOLLO): a randomised, controlled, phase 3 trial. Lancet Oncol. 2025 Jun;26(6):719-731. doi: 10.1016/S1470-2045(25)00190-1. Epub 2025 May 8. PMID 40349716